CLINICAL TRIAL: NCT00481637
Title: Tumor Immunity in Neurologically Normal Patients
Brief Title: Study to Evaluate Immune Responses in Neurologically Normal Cancer Patients
Status: Completed | Type: Observational
Sponsor: Rockefeller University (Other)
Responsible Party: Sponsor
Other Study IDs: RDA-0269
Record Dates: First submitted 2007-06-01; First posted 2007-06-04 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Cancer
Keywords: paraneoplastic; autoimmunity;
MeSH Terms: conditions — Neoplasms; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cancer patients: SCLC and gynecological cancer patients and unrelated cancer patients with presence of PND-specific CTLs.
- Normal: Normal volunteers

SUMMARY:
The purpose of this study is to study whether immune cells capable of killing tumors that express proteins associated with paraneoplastic neurologic syndrome (PNS) can be found in small cell lung cancer and ovarian cancer patients. The presence of these cells may play a role in tumor immunity in these patients. The protocol involves neurological examinations and collection of blood.

DETAILED DESCRIPTION:
See brief description

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ages 25 -75
2. If leukapheresis:

   Hepatitis B surface antigen negative if tested* Hepatitis C antibody negative if tested* HIV antibody negative if tested* Venereal disease reaction level (VDRL) negative if tested* No known IV drug users Hemoglobin > 8.5 White blood cell count > 3,800 Platelets > 120,000 International normalized ratio (INR) < 2 (verified only if clinically indicated)
3. If large blood draw (1/2 to 1 unit) in lieu of leukapheresis:

Hepatitis B surface antigen negative if tested* Hepatitis C antibody negative if tested* HIV antibody negative if tested* VDRL negative if tested* No known IV drug users HgB > 10.0 WBC > 3,800 Platelets > 120,000 INR < 2 (verified only if clinically indicated)

Exclusion Criteria:

No known neurologic disease 2. No known central nervous system (CNS) metastasis on clinical exam 3. No chemotherapy within 1 month 4. No New York Heart Association class III/IV status 5. No pulmonary disease which limits daily activities 6. No anticoagulation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with SCLC and gynecologic (breast or ovarian) tumors and patients with unrelated cancers. Also healthy volunteers will be included as a comparison group in this study.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 1998-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Paraneoplastic neoplastic disease antibody titer, Cytotoxic T Lymphocyte activity, and clinical data in neurologically normal patients with small cell lung cancer and gynecologic tumors, with tumors unrelated to PNDs, and in normal control patients. | Duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Robert Darnell, MD, PHD, Principal Investigator — Rockefeller University
Locations (1):
- Rockefeller University Hospital, New York, New York, United States